CLINICAL TRIAL: NCT00842530
Title: Efficacy and Safety of Dengue Vaccine in Healthy Children Aged 4 to 11 Years in Thailand
Brief Title: Efficacy and Safety of Dengue Vaccine in Healthy Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CYD23; 2014-001710-25 (EudraCT Number)
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Dengue Virus; Dengue Fever; Dengue Hemorrhagic Fever; Dengue Diseases
Keywords: Dengue virus; Dengue fever; Dengue hemorrhagic fever; Dengue diseases; Dengue vaccine
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Dengue Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The observer-blind design was chosen since the products have different appearances and could be recognized. The person who performed vaccinations knew which product was administered while neither the participant nor the Investigator in charge of safety evaluation knew which product was injected. To maintain the blind and minimize the potential bias, the control group used the same route and schedule as the study vaccine.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYD Dengue Vaccine Group (Experimental): Participants (both Cohort 1 and 2) received 3 injections of the CYD Dengue vaccine, 1 injection each at 0, 6, and 12 months.
  Interventions: Biological: CYD Dengue Vaccine
- Control Group (Placebo Comparator): Participants (Cohort 1) received rabies vaccine at Month 0 and placebo at 6 and 12 months. Participants (Cohort 2) received placebo at 0, 6, and 12 months.
  Interventions: Biological: Inactivated rabies virus vaccine; Biological: Placebo

INTERVENTIONS:
Biological: CYD Dengue Vaccine — 0.5 mL, Subcutaneous
  Other Names: Dengvaxia
  Arms: CYD Dengue Vaccine Group
Biological: Inactivated rabies virus vaccine — 0.5 mL, Subcutaneous
  Other Names: Verorab®
  Arms: Control Group
Biological: Placebo — Sodium chloride 0.9%
  Arms: Control Group

SUMMARY:
The primary objective of the study was to assess the efficacy of CYD dengue vaccine after three injections in preventing symptomatic virologically-confirmed dengue (VCD) cases, regardless of the severity, due to any of the four serotypes in children aged 4 to 11 years at the time of inclusion.

Secondary objectives included to assess:

* Vaccine efficacy against severe VCD cases
* Vaccine efficacy against VCD cases following at least two injections with CYD dengue vaccine
* Immune response to CYD dengue vaccine
* Safety profile of CYD dengue vaccine. Safety assessments include solicited reactions within 7 or 14 days after each injection, unsolicited adverse events within 28 days after each injection, and serious adverse events during the study period.

Other objectives included:

* Vaccine efficacy against VCD cases following at least one injection with CYD dengue vaccine
* Vaccine efficacy against VCD cases due to each serotype
* Participants with clinical signs and symptoms for VCD

DETAILED DESCRIPTION:
Participants (both cohort 1 and 2) received 3 injections of CYD dengue vaccine. Participants (Cohort 1) received rabies vaccine at Month 0 and placebo at 6 and 12 months. Participants (cohort 2) received placebo at 0, 6, and 12 months.

Dengue cases were collected for assessment of efficacy during the Active Phase from first injection until at least 13 months after the third injection. A subset of participants were also evaluated for reactogenicity and immunogenicity.

Symptomatic VCD cases were defined as acute febrile illness with fever lasting for at least 1 day (temperature >= 37.5°C measured at least twice with an interval of at least 4 hours), confirmed by reverse transcriptase-polymerase chain reaction and/or dengue non-structural protein 1 (NS1) enzyme-linked immunosorbent assay antigen test, and occurring >28 days after the third injection.

Dengue hemorrhagic fever (DHF) Grade I, II, III, and IV according to the 1999 World Health Organization (WHO) definition:

Clinical Manifestations: a) Fever: acute onset, high and continuous, lasting 2 to 7 days. b) Any of the following hemorrhagic manifestations (including at least a positive tourniquet test): petechiae, purpura, ecchymosis, epistaxis, gum bleeding, and hematemesis and/or melena.

Laboratory Findings: c) thrombocytopenia (platelet count = 100 000/mm3 or less) d) Plasma leakage as shown by hemoconcentration (hematocrit increased by 20% or more) or pleural effusion (seen on chest X-ray) and/or hypoalbuminemia.

DHF was graded as follows: Grade I: Fever accompanied by non-specific constitutional symptoms; the only hemorrhagic manifestation is a positive tourniquet test. Grade II: Spontaneous bleeding in addition to the manifestations of Grade I participants, usually in the form of skin and/or other hemorrhages. Grade III: Circulatory failure manifested by rapid and weak pulse, narrowing of pulse pressure (20 mmHg or less) or hypotension, with the presence of cold clammy skin and restlessness. Grade IV: Profound shock with undetectable blood pressure and pulse.

Independent Data Monitoring Committee (IDMC) severity criteria:- 1) Thrombocytopenia: platelet count ≤ 50 000/mm^3 ; 2) Any hemorrhage that needs blood transfusion; 3) Objective evidence of capillary permeability documented by one or several of the following: a) Increase in hematocrit by >= 20 percent (%) compared to normal for age, or [(Maximum hematocrit - minimum hematocrit)/min]*100% >= 20%, b) Pleural or abdominal (ascites) effusion (diagnosed either by clinical signs or radiography or other imaging method), c) Hypoproteinemia; 4) Signs of circulatory failure manifested by: a) Narrow pulse pressure <20mm Hg, or hypotension for age (as defined by systolic pressure <80 mm Hg in children <5 years and systolic pressure < 90 mm Hg in children >= 5 years), and b) Rapid and weak pulse, and c) Signs of poor capillary perfusion (cold and clammy extremities, delayed capillary refill); 5) Visceral Manifestations such as: a) Neurological symptoms (convulsions or change in level of consciousness), b) Hepatic failure or elevation of hepatic enzyme (>5-fold normal level), c) Metabolic (hypoglycemia) or electrolyte (hyponatremia, hypocalcemia) disturbances or volume overload (acute pulmonary edema or congestive heart failure), d) Other visceral manifestations such as cardiomyopathy, acute renal failure, acute respiratory failure, cholecystitis.

ELIGIBILITY:
Inclusion Criteria :

* Aged 4 to 11 years on the day of inclusion.
* Participant in good health, based on medical history and physical examination.
* Provision of assent form signed by the participants (for participants >= 7 years old) and informed consent form signed by the parent or another legally acceptable representative.
* Participant and parent/ legally acceptable representative able to attend all scheduled visits and to comply with all trial procedures.
* Participant attended one of the schools involved in the trial and living in the Ratchaburi Province.
* For a female participant of child-bearing potential (girls post-menarche), avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to first vaccination, until at least 4 weeks after the last vaccination.

Exclusion Criteria :

* Febrile illness (temperature >= 37.5°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment.
* For a female participant of child-bearing potential (girls post-menarche), known pregnancy or positive urine pregnancy test on the day of the first trial vaccination.
* Personal or family history of thymic pathology (thymoma), thymectomy, or myasthenia.
* Planned participation in another clinical trial during the present trial period.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy, or long-term systemic corticosteroids therapy.
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccines or to a vaccine containing any of the same substances.
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator.
* Receipt of blood or blood-derived products in the past 3 months.
* Participant deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following the first trial vaccination.e
* Participant who plans to attend another school (outside the trial area) or move to another city in the coming 30 months.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4002 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Sanofi Pasteur Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Sabchareon A, Wallace D, Lang J, Bouckenooghe A, Moureau A. Efficacy of tetravalent dengue vaccine in Thai schoolchildren - Authors' reply. Lancet. 2013 Mar 30;381(9872):1094-5. doi: 10.1016/S0140-6736(13)60755-2. No abstract available. PMID 23540847
- [Derived] Forrat R, Dayan GH, DiazGranados CA, Bonaparte M, Laot T, Capeding MR, Sanchez L, Coronel DL, Reynales H, Chansinghakul D, Hadinegoro SRS, Perroud AP, Frago C, Zambrano B, Machabert T, Wu Y, Luedtke A, Price B, Vigne C, Haney O, Savarino SJ, Bouckenooghe A, Noriega F. Analysis of Hospitalized and Severe Dengue Cases Over the 6 years of Follow-up of the Tetravalent Dengue Vaccine (CYD-TDV) Efficacy Trials in Asia and Latin America. Clin Infect Dis. 2021 Sep 15;73(6):1003-1012. doi: 10.1093/cid/ciab288. PMID 33822015
- [Derived] Sridhar S, Luedtke A, Langevin E, Zhu M, Bonaparte M, Machabert T, Savarino S, Zambrano B, Moureau A, Khromava A, Moodie Z, Westling T, Mascarenas C, Frago C, Cortes M, Chansinghakul D, Noriega F, Bouckenooghe A, Chen J, Ng SP, Gilbert PB, Gurunathan S, DiazGranados CA. Effect of Dengue Serostatus on Dengue Vaccine Safety and Efficacy. N Engl J Med. 2018 Jul 26;379(4):327-340. doi: 10.1056/NEJMoa1800820. Epub 2018 Jun 13. PMID 29897841
- [Derived] Plennevaux E, Sabchareon A, Limkittikul K, Chanthavanich P, Sirivichayakul C, Moureau A, Boaz M, Wartel TA, Saville M, Bouckenooghe A. Detection of dengue cases by serological testing in a dengue vaccine efficacy trial: Utility for efficacy evaluation and impact of future vaccine introduction. Vaccine. 2016 May 23;34(24):2707-12. doi: 10.1016/j.vaccine.2016.04.028. Epub 2016 Apr 18. PMID 27102820
- [Derived] Hadinegoro SR, Arredondo-Garcia JL, Capeding MR, Deseda C, Chotpitayasunondh T, Dietze R, Muhammad Ismail HI, Reynales H, Limkittikul K, Rivera-Medina DM, Tran HN, Bouckenooghe A, Chansinghakul D, Cortes M, Fanouillere K, Forrat R, Frago C, Gailhardou S, Jackson N, Noriega F, Plennevaux E, Wartel TA, Zambrano B, Saville M; CYD-TDV Dengue Vaccine Working Group. Efficacy and Long-Term Safety of a Dengue Vaccine in Regions of Endemic Disease. N Engl J Med. 2015 Sep 24;373(13):1195-206. doi: 10.1056/NEJMoa1506223. Epub 2015 Jul 27. PMID 26214039
- [Derived] Sabchareon A, Wallace D, Sirivichayakul C, Limkittikul K, Chanthavanich P, Suvannadabba S, Jiwariyavej V, Dulyachai W, Pengsaa K, Wartel TA, Moureau A, Saville M, Bouckenooghe A, Viviani S, Tornieporth NG, Lang J. Protective efficacy of the recombinant, live-attenuated, CYD tetravalent dengue vaccine in Thai schoolchildren: a randomised, controlled phase 2b trial. Lancet. 2012 Nov 3;380(9853):1559-67. doi: 10.1016/S0140-6736(12)61428-7. Epub 2012 Sep 11. PMID 22975340

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 05 February 2009 to 05 February 2010 at 1 clinical site in Thailand. A total of 4002 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and randomized; however, only 3997 participants received the first vaccination.
Pre-assignment Details: Two-step enrollment approach was followed. Cohort 1 (100 participants [CYD vaccine arm] received CYD vaccine as Injection [Inj.] 1 and 50 [control group arm] received rabies vaccine as Inj. 1) was enrolled first. After 14 days review of Cohort 1 safety data in both arms, cohort 2 was enrolled (2569 participants in CYD group; 1283 in control group).
Groups:
- CYD Dengue Vaccine Group: Participants (both Cohort 1 and 2) received 3 injections of the CYD Dengue vaccine, 1 Inj. each at 0, 6 months, and 12 months.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Group | Control Group
Started | 2669 | 1333
Received Vaccination 1 | 2666 | 1331
Received Vaccination 2 | 2584 | 1300
Received Vaccination 3 | 2557 | 1282
Completed | 2552 | 1276
Not Completed | 117 | 57
Not completed — Serious adverse event | 0 | 6
Not completed — Other adverse event | 6 | 1
Not completed — Protocol Violation | 32 | 14
Not completed — Lost to Follow-up | 6 | 8
Not completed — Withdrawal by Subject | 73 | 28

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who have received at least one injection and were analyzed according to the treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group | Control Group | Total
Number analyzed (Participants) | 2666 | 1331 | 3997
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.16 (2.03) | 8.20 (2.05) | 8.17 (2.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1376 | 696 | 2072
  Male | 1290 | 635 | 1925

OUTCOME MEASURES:

1. Primary Outcome: Number of Symptomatic Virologically-Confirmed Dengue (VCD) Cases During the Active Phase Post-dose 3 Following Inj. With Either CYD Dengue Vaccine or a Placebo
Description: Symptomatic VCD cases were defined as acute febrile illness with fever lasting for at least 1 day (temperature >= 37.5 degree Celsius (°C) measured at least twice with an interval of at least 4 hours), confirmed by reverse transcriptase-polymerase chain reaction and/or dengue non-structural protein-1 (NS1) enzyme-linked immunosorbent assay antigen test, and occurring more than 28 days after the third injection. Vaccine efficacy was reported as density incidence (cases/100 person-years at risk). Density incidence was defined as the number of VCD cases divided by the cumulative person-years at risk.
Time Frame: 28 days Post-Inj. 3 up to the end of Active Phase (up to 13 months Post-Inj. 3, i.e. up to 25 months)
Population: Analysis was performed on Per-protocol analysis (PPA) set for efficacy which included participants with no protocol deviations. Participants with following protocol deviations were excluded: inclusion criteria not met or exclusion criteria met, randomization error, Inj. not performed, code breaking and delay between the inj. not respected.
Measure: Number; unit: Cases
Groups:
- CYD Dengue Vaccine Group: Participants (both Cohort 1 and 2) received 3 injections of the CYD Dengue vaccine, 1 Inj. each at 0, 6, and 12 months.
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2452 | 1221
Cases | 45 | 32
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Control Group; Vaccine efficacy of CYD dengue vaccine: The statistical methodology was based on the use of the two-sided 95% confidence interval (CI) of the vaccine efficacy. The CI was calculated using the exact method conditional on the total number of cases in both groups; Test type: Superiority — The vaccine efficacy of the CYD dengue vaccine against severe VCD cases was considered significant only if the lower bound of its 95% CI was greater than 0%; Vaccine efficacy (%) = 30.2, 95% CI 2-sided [-13.4 to 56.6]

2. Secondary Outcome: Number of Severe VCD Cases During the Active Phase Post-dose 3 Following Inj. With Either CYD Dengue Vaccine or a Placebo
Description: The severity of VCD cases was assessed by WHO 1999 severity assessment and IDMC clinical assessment. Dengue Hemorrhagic Fever (DHF) Grade I, II, III, and IV : Clinical Manifestations: a) Fever: acute onset, high and continuous, lasting 2-7 days, b) Any of hemorrhagic manifestations: petechiae, purpura, ecchymosis, epistaxis, gum bleeding, and hematemesis and/or melena, c) thrombocytopenia (platelet count=100 000/mm3 or less) d) Plasma leakage as shown by hemoconcentration (hematocrit increased by 20% or more) or pleural effusion and/or hypoalbuminemia. IDMC severity criteria: 1) Thrombocytopenia: platelet count <= 50 000/mm^3; 2) Hemorrhage that needs blood transfusion; 3) Objective evidence of capillary permeability 4) Signs of circulatory failure; 5) Visceral Manifestations. Vaccine efficacy was reported as density incidence (cases/100 person-years at risk). Density incidence was defined as the number of VCD cases divided by the cumulative person-years at risk.
Time Frame: 28 days Post-Inj. 3 up to the end of Active Phase (up to 13 months Post-Inj. 3, i.e. up to 25 months)
Population: Analysis was performed on PPA set for efficacy.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2452 | 1221
Cases
  Severe VCD cases (IDMC clinical assessment) | 1 | 2
  Severe VCD cases (WHO 1999 severity assessment) | 2 | 2
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Control Group; Vaccine efficacy against severe VCD (IDMC); Test type: Other — The statistical methodology was based on the use of the two-sided 95% CI of the vaccine efficacy. The CI was calculated using the exact method conditional on the total number of cases in both groups. The vaccine efficacy of the CYD dengue vaccine against severe VCD cases was considered significant if the lower bound of its 95% CI was greater than 0%; Vaccine efficacy (%) = 75.2, 95% CI 2-sided [-377 to 99.6]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Group vs Control Group; Vaccine efficacy of against severe VCD (WHO 1999); Test type: Other — [test comment as in outcome 2, analysis 1]; Vaccine efficacy (%) = 50.3, 95% CI 2-sided [-585 to 96.4]

3. Secondary Outcome: Number of Symptomatic VCD Cases During the Active Phase Following at Least Two Inj. With Either CYD Dengue Vaccine or a Placebo
Description: Symptomatic VCD cases were defined as acute febrile illness with fever lasting for at least 1 day (temperature >= 37.5°C measured at least twice with an interval of at least 4 hours), confirmed by dengue reverse transcriptase-polymerase chain reaction and/or dengue NS1 enzyme-linked immunosorbent assay antigen test, and occurring more than 28 days after the third injection. Vaccine efficacy was reported as density incidence (cases/100 person-years at risk). Density incidence was defined as the number of VCD cases divided by the cumulative person-years at risk.
Time Frame: 28 days Post-Inj. 2 up to Inj. 3, 28 days Post-Inj. 2 up to end of Active Phase ( up to 25 months)
Population: Analysis was performed on Other Efficacy Analysis Set 2 which included all participants who received at least the two first injections.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2584 | 1300
Cases
  Cases: 28 days Post-Inj. 2 up to Inj. 3 | 14 | 12
  Cases:28 days Post-Inj. 2 upto end of Active Phase | 61 | 47
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Control Group; Vaccine efficacy:- 28 days Post-Inj. 2 up to Inj. 3; Test type: Superiority — The statistical methodology was based on the use of the two-sided 95% CI of the vaccine efficacy. The CI was calculated using the exact method conditional on the total number of cases in both groups. The vaccine efficacy of the CYD dengue vaccine against severe VCD cases was considered significant only if the lower bound of its 95% CI was greater than 0%; Vaccine efficacy (%) = 41.5, 95% CI 2-sided [-38.4 to 74.9]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Group vs Control Group; Vaccine efficacy: 28 days Post-Inj. 2 up to end of Active Phase; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Vaccine efficacy (%) = 35.3, 95% CI 2-sided [3.3 to 56.5]

4. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Each Serotype With the Parental Dengue Virus Strain Before and Following Inj. With Either CYD Dengue Vaccine or a Placebo
Description: GMT of antibodies against each serotype with the parental dengue virus strain were assessed by the plaque reduction neutralization test (PRNT).
Time Frame: Pre-Inj. 1, 2, and 3, 28 days Post-Inj. 1, 2 and 3 and 1 year Post-Inj. 3
Population: Analysis was performed on Full Analysis Set for Immunogenicity defined as the participants included in the subgroup for Immunogenicity assessment who have received at least one dose and who had a blood sample drawn after vaccination. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 197 | 99
Titers (1/dilution)
  Dengue Virus Serotype 1; Pre-Inj. 1 | 42.8 [30.7 to 59.6] | 26.6 [17.6 to 40.2]
  Dengue Virus Serotype 1; Post-Inj. 1: number analyzed (Participants) | 197 | 98
  Dengue Virus Serotype 1; Post-Inj. 1 | 94.4 [66.4 to 134] | 27.7 [18.1 to 42.3]
  Dengue Virus Serotype 1; Pre-Inj. 2: number analyzed (Participants) | 188 | 95
  Dengue Virus Serotype 1; Pre-Inj. 2 | 78.0 [54.4 to 112] | 30.5 [19.8 to 47.1]
  Dengue Virus Serotype 1; Post-Inj. 2: number analyzed (Participants) | 189 | 96
  Dengue Virus Serotype 1; Post-Inj. 2 | 184 [137 to 247] | 28.3 [18.2 to 43.8]
  Dengue Virus Serotype 1; Pre-Inj. 3: number analyzed (Participants) | 188 | 95
  Dengue Virus Serotype 1; Pre-Inj. 3 | 116 [84.8 to 160] | 26.4 [17.1 to 40.8]
  Dengue Virus Serotype 1; Post-Inj. 3: number analyzed (Participants) | 188 | 96
  Dengue Virus Serotype 1; Post-Inj. 3 | 155 [116 to 207] | 27.8 [18.3 to 42.2]
  Dengue Virus Serotype 1; 1 year Post-Inj. 3: number analyzed (Participants) | 187 | 94
  Dengue Virus Serotype 1; 1 year Post-Inj. 3 | 120 [87.0 to 166] | 35.8 [23.1 to 55.4]
  Dengue Virus Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 197 | 98
  Dengue Virus Serotype 2; Pre-Inj. 1 | 56.8 [40.3 to 80.1] | 43.7 [27.8 to 68.7]
  Dengue Virus Serotype 2; Post-Inj. 1 | 195 [143 to 266] | 42.9 [27.2 to 67.6]
  Dengue Virus Serotype 2; Pre-Inj. 2: number analyzed (Participants) | 189 | 96
  Dengue Virus Serotype 2; Pre-Inj. 2 | 152 [109 to 210] | 50.5 [31.9 to 79.9]
  Dengue Virus Serotype 2; Post-Inj. 2: number analyzed (Participants) | 189 | 96
  Dengue Virus Serotype 2; Post-Inj. 2 | 351 [274 to 449] | 44.6 [28.5 to 69.8]
  Dengue Virus Serotype 2; Pre-Inj. 3: number analyzed (Participants) | 188 | 95
  Dengue Virus Serotype 2; Pre-Inj. 3 | 239 [184 to 311] | 54.8 [34.3 to 87.4]
  Dengue Virus Serotype 2; Post-Inj. 3: number analyzed (Participants) | 188 | 96
  Dengue Virus Serotype 2; Post-Inj. 3 | 358 [283 to 453] | 52.2 [32.3 to 84.4]
  Dengue Virus Serotype 2; 1 year Post-Inj. 3: number analyzed (Participants) | 187 | 94
  Dengue Virus Serotype 2; 1 year Post-Inj. 3 | 158 [117 to 213] | 46.1 [29.4 to 72.4]
  Dengue Virus Serotype 3; Pre-Inj. 1 | 31.5 [24.2 to 41.0] | 28.7 [19.3 to 42.6]
  Dengue Virus Serotype 3; Post-Inj. 1 | 112 [85.8 to 146] | 27.0 [18.3 to 39.8]
  Dengue Virus Serotype 3; Pre-Inj. 2: number analyzed (Participants) | 189 | 95
  Dengue Virus Serotype 3; Pre-Inj. 2 | 81.3 [61.6 to 107] | 31.1 [20.6 to 46.9]
  Dengue Virus Serotype 3; Post-Inj. 2: number analyzed (Participants) | 189 | 96
  Dengue Virus Serotype 3; Post-Inj. 2 | 218 [178 to 267] | 26.9 [18.2 to 39.8]
  Dengue Virus Serotype 3; Pre-Inj. 3: number analyzed (Participants) | 188 | 95
  Dengue Virus Serotype 3; Pre-Inj. 3 | 240 [193 to 299] | 50.3 [32.1 to 78.9]
  Dengue Virus Serotype 3; Post-Inj. 3: number analyzed (Participants) | 188 | 96
  Dengue Virus Serotype 3; Post-Inj. 3 | 351 [289 to 428] | 46.2 [29.9 to 71.4]
  Dengue Virus Serotype 3; 1 year Post-Inj. 3: number analyzed (Participants) | 187 | 94
  Dengue Virus Serotype 3; 1 year Post-Inj. 3 | 125 [97.2 to 161] | 35.1 [23.0 to 53.6]
  Dengue Virus Serotype 4; Pre-Inj. 1 | 28.1 [21.7 to 36.4] | 23.2 [15.6 to 34.6]
  Dengue Virus Serotype 4; Post-Inj. 1 | 138 [106 to 178] | 24.2 [16.4 to 35.8]
  Dengue Virus Serotype 4; Pre-Inj. 2: number analyzed (Participants) | 189 | 95
  Dengue Virus Serotype 4; Pre-Inj. 2 | 74.0 [57.2 to 95.7] | 25.6 [16.9 to 38.8]
  Dengue Virus Serotype 4; Post-Inj. 2: number analyzed (Participants) | 189 | 96
  Dengue Virus Serotype 4; Post-Inj. 2 | 183 [151 to 220] | 25.3 [17.0 to 37.5]
  Dengue Virus Serotype 4; Pre-Inj. 3: number analyzed (Participants) | 188 | 95
  Dengue Virus Serotype 4; Pre-Inj. 3 | 110 [89.3 to 136] | 24.4 [16.7 to 35.8]
  Dengue Virus Serotype 4; Post-Inj. 3: number analyzed (Participants) | 188 | 96
  Dengue Virus Serotype 4; Post-Inj. 3 | 151 [128 to 178] | 22.1 [15.3 to 32.0]
  Dengue Virus Serotype 4; 1 year Post-Inj. 3: number analyzed (Participants) | 187 | 94
  Dengue Virus Serotype 4; 1 year Post-Inj. 3 | 152 [120 to 192] | 45.9 [30.4 to 69.3]

5. Secondary Outcome: GMTs of Antibodies Against Each Serotype With the Parental Dengue Virus Strain in Dengue-Immune Participants Before and Following Inj. With Either CYD Dengue Vaccine or a Placebo
Description: GMTs of antibodies against each serotype with the parental dengue virus strain were assessed by the PRNT. Dengue immune participants were defined as those participants with titers >= 10 (1/dilution) against at least one dengue serotype at baseline.
Time Frame: Pre-Inj. 1, 2, and 3, 28 days Post-Inj. 1, 2 and 3 and 1 year Post-Inj. 3
Population: Analysis was performed on Full Analysis Set for Immunogenicity. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 138 | 68
Titers (1/dilution)
  Dengue Virus Serotype 1; Pre-Inj. 1 | 107 [73.1 to 157] | 57.0 [34.3 to 94.7]
  Dengue Virus Serotype 1; Post-Inj. 1: number analyzed (Participants) | 138 | 67
  Dengue Virus Serotype 1; Post-Inj. 1 | 235 [158 to 349] | 59.7 [35.3 to 101]
  Dengue Virus Serotype 1; Pre-Inj. 2: number analyzed (Participants) | 133 | 65
  Dengue Virus Serotype 1; Pre-Inj. 2 | 193 [130 to 287] | 68.4 [40.4 to 116]
  Dengue Virus Serotype 1; Post-Inj. 2: number analyzed (Participants) | 134 | 66
  Dengue Virus Serotype 1; Post-Inj. 2 | 371 [269 to 511] | 58.9 [34.0 to 102]
  Dengue Virus Serotype 1; Pre-Inj. 3: number analyzed (Participants) | 133 | 65
  Dengue Virus Serotype 1; Pre-Inj. 3 | 254 [180 to 360] | 49.3 [28.2 to 86.1]
  Dengue Virus Serotype 1; Post-Inj. 3: number analyzed (Participants) | 133 | 66
  Dengue Virus Serotype 1; Post-Inj. 3 | 283 [202 to 397] | 50.6 [29.8 to 85.6]
  Dengue Virus Serotype 1; 1 year Post-Inj. 3: number analyzed (Participants) | 133 | 65
  Dengue Virus Serotype 1; 1 year Post-Inj. 3 | 262 [185 to 371] | 67.0 [39.9 to 113]
  Dengue Virus Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 138 | 67
  Dengue Virus Serotype 2; Pre-Inj. 1 | 161 [111 to 233] | 119 [72.3 to 197]
  Dengue Virus Serotype 2; Post-Inj. 1 | 449 [324 to 623] | 112 [67.0 to 188]
  Dengue Virus Serotype 2; Pre-Inj. 2: number analyzed (Participants) | 134 | 66
  Dengue Virus Serotype 2; Pre-Inj. 2 | 340 [240 to 481] | 139 [84.8 to 229]
  Dengue Virus Serotype 2; Post-Inj. 2: number analyzed (Participants) | 134 | 66
  Dengue Virus Serotype 2; Post-Inj. 2 | 619 [471 to 813] | 117 [71.2 to 191]
  Dengue Virus Serotype 2; Pre-Inj. 3: number analyzed (Participants) | 133 | 65
  Dengue Virus Serotype 2; Pre-Inj. 3 | 413 [308 to 555] | 132 [78.4 to 223]
  Dengue Virus Serotype 2; Post-Inj. 3: number analyzed (Participants) | 133 | 66
  Dengue Virus Serotype 2; Post-Inj. 3 | 562 [427 to 741] | 118 [68.0 to 206]
  Dengue Virus Serotype 2; 1 year Post-Inj. 3: number analyzed (Participants) | 133 | 65
  Dengue Virus Serotype 2; 1 year Post-Inj. 3 | 332 [246 to 450] | 99.1 [59.5 to 165]
  Dengue Virus Serotype 3; Pre-Inj. 1 | 69.2 [51.8 to 92.5] | 63.7 [40.1 to 101]
  Dengue Virus Serotype 3; Post-Inj. 1 | 216 [163 to 287] | 56.1 [35.2 to 89.5]
  Dengue Virus Serotype 3; Pre-Inj. 2: number analyzed (Participants) | 134 | 65
  Dengue Virus Serotype 3; Pre-Inj. 2 | 152 [113 to 205] | 66.1 [40.2 to 109]
  Dengue Virus Serotype 3; Post-Inj. 2: number analyzed (Participants) | 134 | 66
  Dengue Virus Serotype 3; Post-Inj. 2 | 308 [245 to 389] | 52.3 [32.3 to 84.6]
  Dengue Virus Serotype 3; Pre-Inj. 3: number analyzed (Participants) | 133 | 65
  Dengue Virus Serotype 3; Pre-Inj. 3 | 361 [285 to 457] | 107 [64.7 to 178]
  Dengue Virus Serotype 3; Post-Inj. 3: number analyzed (Participants) | 133 | 66
  Dengue Virus Serotype 3; Post-Inj. 3 | 469 [368 to 599] | 91.7 [55.7 to 151]
  Dengue Virus Serotype 3; 1 year Post-Inj. 3: number analyzed (Participants) | 133 | 65
  Dengue Virus Serotype 3; 1 year Post-Inj. 3 | 213 [162 to 280] | 61.8 [37.7 to 101]
  Dengue Virus Serotype 4; Pre-Inj. 1 | 58.8 [43.9 to 78.7] | 46.8 [28.3 to 77.2]
  Dengue Virus Serotype 4; Post-Inj. 1 | 212 [162 to 277] | 49.7 [30.7 to 80.5]
  Dengue Virus Serotype 4; Pre-Inj. 2: number analyzed (Participants) | 134 | 65
  Dengue Virus Serotype 4; Pre-Inj. 2 | 121 [90.5 to 163] | 53.2 [31.7 to 89.3]
  Dengue Virus Serotype 4; Post-Inj. 2: number analyzed (Participants) | 134 | 66
  Dengue Virus Serotype 4; Post-Inj. 2 | 266 [216 to 327] | 51.8 [32.0 to 84.0]
  Dengue Virus Serotype 4; Pre-Inj. 3: number analyzed (Participants) | 133 | 65
  Dengue Virus Serotype 4; Pre-Inj. 3 | 170 [137 to 212] | 45.3 [28.3 to 72.6]
  Dengue Virus Serotype 4; Post-Inj. 3: number analyzed (Participants) | 133 | 66
  Dengue Virus Serotype 4; Post-Inj. 3 | 198 [164 to 239] | 40.1 [25.3 to 63.3]
  Dengue Virus Serotype 4; 1 year Post-Inj. 3: number analyzed (Participants) | 133 | 65
  Dengue Virus Serotype 4; 1 year Post-Inj. 3 | 234 [179 to 305] | 89.6 [56.0 to 143]

6. Secondary Outcome: GMTs of Antibodies Against Each Serotype With the Parental Dengue Virus Strain in Dengue Non-Immune Participants Before and Following Inj. With Either CYD Dengue Vaccine or a Placebo
Description: GMTs of antibodies against each serotype with the parental dengue virus strain were assessed by the PRNT. Dengue non-immune participants were defined as participants with titers < 10 (1/dilution) against all four dengue serotypes at baseline.
Time Frame: Pre-Inj. 1, 2, and 3, 28 days Post-Inj. 1, 2 and 3 and 1 year Post-Inj. 3
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 59 | 31
Titers (1/dilution)
  Dengue Virus Serotype 1; Pre-Inj. 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Dengue Virus Serotype 1; Post-Inj. 1 | 11.2 [8.04 to 15.5] | 5.24 [4.76 to 5.76]
  Dengue Virus Serotype 1; Pre-Inj. 2: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 1; Pre-Inj. 2 | 8.72 [6.07 to 12.5] | 5.31 [4.87 to 5.80]
  Dengue Virus Serotype 1; Post-Inj. 2: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 1; Post-Inj. 2 | 33.3 [22.7 to 49.0] | 5.62 [4.76 to 6.64]
  Dengue Virus Serotype 1; Pre-Inj. 3: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 1; Pre-Inj. 3 | 17.6 [12.3 to 25.3] | 6.86 [4.89 to 9.61]
  Dengue Virus Serotype 1; Post-Inj. 3: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 1; Post-Inj. 3 | 35.8 [25.4 to 50.5] | 7.47 [5.18 to 10.8]
  Dengue Virus Serotype 1; 1 year Post-Inj. 3: number analyzed (Participants) | 54 | 29
  Dengue Virus Serotype 1; 1 year Post-Inj. 3 | 17.6 [12.0 to 25.8] | 8.76 [5.01 to 15.3]
  Dengue Virus Serotype 2; Pre-Inj. 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Dengue Virus Serotype 2; Post-Inj. 1 | 27.7 [18.6 to 41.1] | 5.19 [4.81 to 5.60]
  Dengue Virus Serotype 2; Pre-Inj. 2: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 2; Pre-Inj. 2 | 21.3 [14.1 to 32.1] | 5.41 [4.83 to 6.05]
  Dengue Virus Serotype 2; Post-Inj. 2: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 2; Post-Inj. 2 | 88.3 [65.3 to 119] | 5.38 [4.63 to 6.26]
  Dengue Virus Serotype 2; Pre-Inj. 3: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 2; Pre-Inj. 3 | 63.7 [43.8 to 92.5] | 8.12 [4.93 to 13.4]
  Dengue Virus Serotype 2; Post-Inj. 3: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 2; Post-Inj. 3 | 120 [89.7 to 162] | 8.64 [4.96 to 15.0]
  Dengue Virus Serotype 2; 1 year Post-Inj. 3: number analyzed (Participants) | 54 | 29
  Dengue Virus Serotype 2; 1 year Post-Inj. 3 | 25.2 [16.1 to 39.4] | 8.31 [4.85 to 14.2]
  Dengue Virus Serotype 3; Pre-Inj. 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Dengue Virus Serotype 3; Post-Inj. 1 | 23.9 [16.6 to 34.4] | 5.43 [4.59 to 6.42]
  Dengue Virus Serotype 3; Pre-Inj. 2: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 3; Pre-Inj. 2 | 17.7 [11.8 to 26.5] | 6.05 [5.00 to 7.33]
  Dengue Virus Serotype 3; Post-Inj. 2: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 3; Post-Inj. 2 | 93.6 [68.7 to 128] | 6.23 [4.94 to 7.85]
  Dengue Virus Serotype 3; Pre-Inj. 3: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 3; Pre-Inj. 3 | 89.3 [61.3 to 130] | 9.78 [5.41 to 17.7]
  Dengue Virus Serotype 3; Post-Inj. 3: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 3; Post-Inj. 3 | 174 [137 to 223] | 10.2 [5.67 to 18.3]
  Dengue Virus Serotype 3; 1 year Post-Inj. 3: number analyzed (Participants) | 54 | 29
  Dengue Virus Serotype 3; 1 year Post-Inj. 3 | 33.9 [23.2 to 49.5] | 9.89 [5.35 to 18.3]
  Dengue Virus Serotype 4; Pre-Inj. 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Dengue Virus Serotype 4; Post-Inj. 1 | 50.0 [29.6 to 84.4] | 5.00 [5.00 to 5.00]
  Dengue Virus Serotype 4; Pre-Inj. 2: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 4; Pre-Inj. 2 | 22.2 [15.3 to 32.2] | 5.26 [4.74 to 5.84]
  Dengue Virus Serotype 4; Post-Inj. 2: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 4; Post-Inj. 2 | 73.0 [55.1 to 96.8] | 5.20 [4.80 to 5.63]
  Dengue Virus Serotype 4; Pre-Inj. 3: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 4; Pre-Inj. 3 | 38.8 [26.5 to 56.7] | 6.41 [4.66 to 8.82]
  Dengue Virus Serotype 4; Post-Inj. 3: number analyzed (Participants) | 55 | 30
  Dengue Virus Serotype 4; Post-Inj. 3 | 78.1 [59.7 to 102] | 5.98 [4.64 to 7.71]
  Dengue Virus Serotype 4; 1 year Post-Inj. 3: number analyzed (Participants) | 54 | 29
  Dengue Virus Serotype 4; 1 year Post-Inj. 3 | 52.3 [36.7 to 74.5] | 10.3 [6.11 to 17.2]

7. Secondary Outcome: Percentage of Participants With Solicited Inj. Site Reactions Following Any and Each Inj. With Either CYD Dengue Vaccine or a Placebo
Description: Solicited Inj. site reactions: Pain, Erythema, and Swelling. Pain: - Grade 1: easily tolerated, Grade 2: sufficiently discomforting to interfere with normal behavior or activities, Grade 3: incapacitating, unable to perform usual activities. Erythema and Swelling: - Grade 1: > 0.0 to < 2.5 cm, Grade 2: >= 2.5 to < 5 cm, Grade 3: >= 5 cm.
Time Frame: 7 days post-any Inj. and each of the 3 Inj.
Population: Analysis was performed in the Reactogenicity Analysis Set, which included all participants who received at least one injection and were considered evaluable for reactogenicity. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 697 | 350
Percentage of participants
  Inj. site Pain; Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Inj. site Pain; Post-Any Inj. | 57.7 | 57.6
  Grade 3 Inj. site Pain; Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Grade 3 Inj. site Pain; Post-Any Inj. | 0.1 | 0.0
  Inj. site Erythema; Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Inj. site Erythema; Post-Any Inj. | 28.6 | 30.7
  Grade 3 Inj. site Erythema; Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Grade 3 Inj. site Erythema; Post-Any Inj. | 0.0 | 0.0
  Inj. site Swelling; Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Inj. site Swelling; Post-Any Inj. | 21.4 | 22.1
  Grade 3 Inj. site Swelling; Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Grade 3 Inj. site Swelling; Post-Any Inj. | 0.3 | 0.3
  Inj. site Pain; Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Inj. site Pain; Post-Inj. 1 | 33.5 | 30.9
  Grade 3 Inj. site Pain; Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Grade 3 Inj. site Pain; Post-Inj. 1 | 0.0 | 0.0
  Inj. site Erythema; Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Inj. site Erythema; Post-Inj. 1 | 13.3 | 16.3
  Grade 3 Inj. site Erythema; Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Grade 3 Inj. site Erythema; Post-Inj. 1 | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Inj. site Swelling; Post-Inj. 1 | 9.0 | 9.2
  Grade 3 Inj. site Swelling; Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Grade 3 Inj. site Swelling; Post-Inj. 1 | 0.3 | 0.3
  Inj. site Pain; Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Inj. site Pain; Post-Inj. 2 | 35.0 | 32.2
  Grade 3 Inj. site Pain; Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Grade 3 Inj. site Pain; Post-Inj. 2 | 0.1 | 0.0
  Inj. site Erythema; Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Inj. site Erythema; Post-Inj. 2 | 13.0 | 14.6
  Grade 3 Inj. site Erythema; Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Grade 3 Inj. site Erythema; Post-Inj. 2 | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Inj. site Swelling; Post-Inj. 2 | 11.1 | 11.1
  Grade 3 Inj. site Swelling; Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Grade 3 Inj. site Swelling; Post-Inj. 2 | 0.0 | 0.0
  Inj. site Pain; Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Inj. site Pain; Post-Inj. 3 | 33.0 | 30.5
  Grade 3 Inj. site Pain; Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Grade 3 Inj. site Pain; Post-Inj. 3 | 0.0 | 0.0
  Inj. site Erythema; Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Inj. site Erythema; Post-Inj. 3 | 13.7 | 14.5
  Grade 3 Inj. site Erythema; Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Grade 3 Inj. site Erythema; Post-Inj. 3 | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Inj. site Swelling; Post-Inj. 3 | 10.4 | 10.9
  Grade 3 Inj. site Swelling; Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Grade 3 Inj. site Swelling; Post-Inj. 3 | 0.0 | 0.0

8. Secondary Outcome: Percentage of Participants With Solicited Systemic Reactions Following Any and Each Inj. With Either CYD Dengue Vaccine or a Placebo
Description: Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Fever:- Grade 1: >=37.5°C to <=38.0°C, Grade 2: >38.0°C to <=39.0°C, Grade 3: >39.0°C. Headache, malaise, myalgia and asthenia: - Grade 1: noticeable but does not interfere with daily activities, Grade 2: interferes with daily activities, Grade 3: prevents daily activities.
Time Frame: 14 days post-any Inj. and each of the 3 Inj.
Population: Analysis was performed on Reactogenicity Analysis Set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 697 | 350
Percentage of participants
  Fever: Post-Any Inj.: number analyzed (Participants) | 692 | 350
  Fever: Post-Any Inj. | 32.2 | 34.3
  Grade 3 Fever: Post-Any Inj.: number analyzed (Participants) | 692 | 350
  Grade 3 Fever: Post-Any Inj. | 1.9 | 4.0
  Headache: Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Headache: Post-Any Inj. | 60.0 | 59.3
  Grade 3 Headache: Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Grade 3 Headache: Post-Any Inj. | 2.2 | 2.6
  Malaise: Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Malaise: Post-Any Inj. | 53.6 | 50.7
  Grade 3 Malaise: Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Grade 3 Malaise: Post-Any Inj. | 1.6 | 2.3
  Myalgia: Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Myalgia: Post-Any Inj. | 50.3 | 47.0
  Grade 3 Myalgia: Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Grade 3 Myalgia: Post-Any Inj. | 1.2 | 2.9
  Asthenia: Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Asthenia: Post-Any Inj. | 43.5 | 41.8
  Grade 3 Asthenia: Post-Any Inj.: number analyzed (Participants) | 692 | 349
  Grade 3 Asthenia: Post-Any Inj. | 1.2 | 2.6
  Fever: Post-Inj. 1: number analyzed (Participants) | 672 | 339
  Fever: Post-Inj. 1 | 13.8 | 14.7
  Grade 3 Fever: Post-Inj. 1: number analyzed (Participants) | 672 | 339
  Grade 3 Fever: Post-Inj. 1 | 1.3 | 1.8
  Headache: Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Headache: Post-Inj. 1 | 39.6 | 35.2
  Grade 3 Headache: Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Grade 3 Headache: Post-Inj. 1 | 1.3 | 1.7
  Malaise: Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Malaise: Post-Inj. 1 | 32.4 | 29.5
  Grade 3 Malaise: Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Grade 3 Malaise: Post-Inj. 1 | 0.9 | 1.1
  Myalgia: Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Myalgia: Post-Inj. 1 | 30.2 | 24.9
  Grade 3 Myalgia: Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Grade 3 Myalgia: Post-Inj. 1 | 0.4 | 2.0
  Asthenia: Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Asthenia: Post-Inj. 1 | 25.3 | 23.5
  Grade 3 Asthenia: Post-Inj. 1: number analyzed (Participants) | 692 | 349
  Grade 3 Asthenia: Post-Inj. 1 | 0.6 | 1.1
  Fever: Post-Inj. 2: number analyzed (Participants) | 654 | 329
  Fever: Post-Inj. 2 | 14.5 | 16.7
  Grade 3 Fever: Post-Inj. 2: number analyzed (Participants) | 654 | 329
  Grade 3 Fever: Post-Inj. 2 | 0.5 | 1.2
  Headache: Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Headache: Post-Inj. 2 | 31.1 | 29.8
  Grade 3 Headache: Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Grade 3 Headache: Post-Inj. 2 | 0.6 | 0.3
  Malaise: Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Malaise: Post-Inj. 2 | 27.7 | 24.9
  Grade 3 Malaise: Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Grade 3 Malaise: Post-Inj. 2 | 0.7 | 0.6
  Myalgia: Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Myalgia: Post-Inj. 2 | 28.6 | 25.1
  Grade 3 Myalgia: Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Grade 3 Myalgia: Post-Inj. 2 | 0.3 | 0.6
  Asthenia: Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Asthenia: Post-Inj. 2 | 21.7 | 21.3
  Grade 3 Asthenia: Post-Inj. 2: number analyzed (Participants) | 668 | 342
  Grade 3 Asthenia: Post-Inj. 2 | 0.4 | 0.3
  Fever: Post-Inj. 3: number analyzed (Participants) | 653 | 334
  Fever: Post-Inj. 3 | 11.3 | 12.9
  Grade 3 Fever: Post-Inj. 3: number analyzed (Participants) | 653 | 334
  Grade 3 Fever: Post-Inj. 3 | 0.2 | 1.5
  Headache: Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Headache: Post-Inj. 3 | 27.0 | 32.5
  Grade 3 Headache: Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Grade 3 Headache: Post-Inj. 3 | 0.6 | 0.9
  Malaise: Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Malaise: Post-Inj. 3 | 25.3 | 24.3
  Grade 3 Malaise: Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Grade 3 Malaise: Post-Inj. 3 | 0.2 | 0.9
  Myalgia: Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Myalgia: Post-Inj. 3 | 26.4 | 24.9
  Grade 3 Myalgia: Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Grade 3 Myalgia: Post-Inj. 3 | 0.5 | 0.3
  Asthenia: Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Asthenia: Post-Inj. 3 | 19.9 | 23.4
  Grade 3 Asthenia: Post-Inj. 3: number analyzed (Participants) | 664 | 338
  Grade 3 Asthenia: Post-Inj. 3 | 0.2 | 1.2

9. Other Pre Specified Outcome: Number of Symptomatic VCD Cases During the Active Phase Following at Least One Inj. With Either CYD Dengue Vaccine or a Placebo
Description: Symptomatic VCD cases were defined as acute febrile illness with fever lasting for at least 1 day (temperature >=37.5°C measured at least twice with an interval of at least 4 hours), confirmed by reverse transcriptase-polymerase chain reaction and/or dengue NS1 enzyme-linked immunosorbent assay antigen test, and occurring more than 28 days after the third injection. Vaccine efficacy was reported as density incidence (cases/100 person-years at risk). Density incidence was defined as the number of VCD cases divided by the cumulative person-years at risk.
Time Frame: Day 0 (Post-Inj.) up to end of Active phase (up to 25 months); 28 days post-Inj. 1 up to end of Active phase (up to 25 months)
Population: Analysis was performed on Other Efficacy Analysis Set 1 which included participants who received at least the first injection.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2666 | 1331
Cases
  Cases:28 days Post-Inj.1 upto end of Active Phase | 75 | 56
  Cases:Day 0 upto end of Active Phase | 76 | 58
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Control Group; Vaccine efficacy: 28 days Post-Inj. 1 up to end of Active Phase; Test type: Other — [test comment as in outcome 2, analysis 1]; Vaccine efficacy (%) = 33.4, 95% CI 2-sided [4.1 to 53.5]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Group vs Control Group; Vaccine efficacy: Day 0 up to end of Active Phase; Test type: Other — [test comment as in outcome 2, analysis 1]; Vaccine efficacy (%) = 34.9, 95% CI 2-sided [6.7 to 54.3]

10. Other Pre Specified Outcome: Number of Participants With One VCD Episode During the Active Phase Due to Each Serotypes Following Inj. With Either CYD Dengue Vaccine or a Placebo
Description: Symptomatic VCD cases were defined as acute febrile illness with fever lasting for at least 1 day (temperature >= 37.5°C measured at least twice with an interval of at least 4 hours), confirmed by reverse transcriptase-polymerase chain reaction and/or dengue NS1 enzyme-linked immunosorbent assay antigen test, and occurring more than 28 days after the third injection. VCD cases confirmed only by NS1 method were classified in the Not Identified category. Cases were defined as the number of participants with at least one symptomatic VCD episode more than 28 days after Inj. 3 (during the Active Phase).
Time Frame: After 28 days Post Inj. 3 up to the end of Active Phase (up to 25 months)
Population: Analysis was performed on Other Efficacy Analysis Set 1.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2666 | 1331
Participants
  Dengue Virus Serotype 1 | 14 | 18
  Dengue Virus Serotype 2 | 52 | 27
  Dengue Virus Serotype 3 | 4 | 11
  Dengue Virus Serotype 4 | 1 | 5
  Not Identified | 5 | 1

11. Other Pre Specified Outcome: Mean Number of Days for Clinical Signs and Symptoms (Fever, Clinical Syndrome and Hospitalization) of VCD During the Active Phase Following Inj. With Either CYD Dengue Vaccine or a Placebo
Description: Clinical signs and symptoms for VCD included the following: fever, clinical syndrome and hospitalization. Duration of each symptom (in days) is reported in this outcome measure.
Time Frame: Day 0 (Post-Inj.) up to end of Active Phase (up to 25 months)
Population: Analysis was performed on Safety Analysis Set. Here, 'overall number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 76 | 62
Days
  Fever | 4.13 (1.98) | 4.40 (1.97)
  Clinical syndrome | 5.39 (2.34) | 5.84 (2.68)
  Hospitalization | 4.91 (1.33) | 5.17 (1.97)

12. Other Pre Specified Outcome: Number of Participants Requiring Hospitalization for VCD During the Active Phase Following Inj. With Either CYD Dengue Vaccine or a Placebo
Time Frame: Day 0 (Post-Inj.) up to end of Active Phase (up to 25 months)
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 76 | 62
participants
  Hospitalization; No | 44 | 32
  Hospitalization; Yes | 32 | 30

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to 13 months Post-Inj. 3 (up to 25 months).
Description: All the vaccinated participants were assessed for SAE during the trial. Non-serious adverse events included solicited injection-site (within 7 days after injection) and solicited systemic reactions (within 14 days after injection), as well as unsolicited non-serious adverse events (within 28 days after injection). These events were assessed in a subset of participants from each group, who had received at least 1 injection.
Arm/Group | CYD Dengue Vaccine Group | Control Group
All-Cause Mortality (participants affected / at risk) | 1/2666 | 4/1331
Serious Adverse Events (participants affected / at risk) | 315/2666 | 176/1331
Other Adverse Events (participants affected / at risk) | 415/697 | 207/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CYD Dengue Vaccine Group (N=2666) | Control Group (N=1331)
Tonsillectomy (Surgical and medical procedures) | 2 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Allergy to arthropod sting (Immune system disorders) | 2 | 3
Perineal laceration (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Chest pain (General disorders) | 0 | 1
Drowning (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 2
Balanitis (Reproductive system and breast disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Vaginal perforation (Reproductive system and breast disorders) | 0 | 1
Accidental exposure (Injury, poisoning and procedural complications) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1
Blast injury (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0
Epiphyseal injury (Injury, poisoning and procedural complications) | 2 | 1
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 2 | 1
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 3
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2
Snake bite (Injury, poisoning and procedural complications) | 5 | 2
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vulva injury (Injury, poisoning and procedural complications) | 1 | 2
Wound (Injury, poisoning and procedural complications) | 3 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 5 | 5
Convulsion (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Febrile convulsion (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Appendicitis perforated (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Food poisoning (Gastrointestinal disorders) | 5 | 1
Gastritis (Gastrointestinal disorders) | 45 | 22
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Mouth cyst (Gastrointestinal disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 1
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 3 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 | 1
Abscess limb (Infections and infestations) | 3 | 0
Abscess of eyelid (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 1
Acute tonsillitis (Infections and infestations) | 8 | 2
Appendicitis (Infections and infestations) | 8 | 4
Arthritis bacterial (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 28 | 14
Bronchitis viral (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 5 | 4
Cellulitis of male external genital (Infections and infestations) | 2 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 19 | 19
Diarrhoea infectious (Infections and infestations) | 8 | 5
Dysentery (Infections and infestations) | 0 | 1
Exanthema subitum (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 44 | 20
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 4 | 5
Lobar pneumonia (Infections and infestations) | 0 | 1
Malaria (Infections and infestations) | 1 | 0
Mumps (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 2
Orchitis (Infections and infestations) | 1 | 1
Otitis media acute (Infections and infestations) | 1 | 2
Perianal abscess (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 44 | 18
Pharyngotonsillitis (Infections and infestations) | 8 | 8
Pneumonia (Infections and infestations) | 3 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pyoderma (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tonsillitis (Infections and infestations) | 3 | 3
Typhus (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Varicella (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 9 | 7
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Viral myositis (Infections and infestations) | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | CYD Dengue Vaccine Group (N=697) | Control Group (N=350)
Headache; Post-Any Injection (Nervous system disorders) | 415/692 | 207/349
Injection site Pain; Post-Any (General disorders) | 399/692 | 201/349
Injection site Erythema; Post-Any Injection (General disorders) | 198/692 | 107/349
Injection site Swelling; Post-Any Injection (General disorders) | 148/692 | 77/349
Fever; Post-Any Injection (General disorders) | 223/692 | 120
Malaise; Post-Any Injection (General disorders) | 371/692 | 177/349
Asthenia; Post-Any Injection (General disorders) | 301/692 | 146/349
Myalgia; Post-Any Injection (Musculoskeletal and connective tissue disorders) | 348/692 | 164/349
Nasopharyngitis (Infections and infestations) | 37 | 18
Pharyngitis (Infections and infestations) | 61 | 32
Upper respiratory tract infection (Infections and infestations) | 78 | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications